CLINICAL TRIAL: NCT02731677
Title: Acupuncture as Adjuvant Therapy for Sleep Disorders in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, NADJA MARIA JORGE ASANO, PRINCIPAL INVESTIGATOR, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE 49662915.4.0000.5208
Record Dates: First submitted 2016-03-22; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Acupuncture was applied on the acupoints F3 - BP6- VB34- IG4 - TA5 - C7 - PC6 - IG11 - VB20 - XIAOCHANXUE, once a week, eight sessions in the experimental group.
  Interventions: Other: Acupuncture
- Control (No Intervention): The control group no suffered intervention.

INTERVENTIONS:
Other: Acupuncture — Acupuncture was applied on the acupoints F3 - BP6- VB34- IG4 - TA5 - C7 - PC6 - IG11 - VB20 - XIAOCHANXUE, once a week, eight sessions in the experimental group.
  Arms: Experimental

SUMMARY:
Sleep disorders correspond to a non-motor symptom present in DP, being represented by daytime sleepiness and maintenance insomnia. This study aims to evaluate the effects of acupuncture on sleep disorders in patients with PD assisted by Pró-Parkinson Program at University Hospital of Pernambuco, Brazil. Its a randomized clinical trial approved by the Ethics Committee for Research with Human. It was included patients with diagnosed with Idiopathic Parkinson's disease, Mini Mental State Examination (MMEE) according to education, stages 1, 2 and 3 in the Hoehn-Yahr scale. It was used the sleep Scale for Parkinson's disease (PDSS), a self-administered scale designed to assess nighttime sleep problems, sleep disorders and excessive daytime sleep. Twenty-two subjects were allocated in two groups: experimental and control. Acupuncture was applied on the acupoints F3 - BP6- VB34- IG4 - TA5 - C7 - PC6 - IG11 - VB20 - XIAOCHANXUE once a week, eight sessions in the experimental group. The control group no suffered intervention. The paired analyzes were performed using the Wilcoxon test and the independent analyzes using the Mann-Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Idiopathic Parkinson's disease
* Mini Mental State Examination (MMSE) According to education
* Stages 1, 2 and 3 in the Hoehn-Yahr scale.

Exclusion Criteria:

* Patients who have another neurological disorder associated with Parkinson's disease
* Cardiac with pacemaker (contraindicated the use of electrotherapy).

Ages: 38 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Scale for Parkinson's disease (PDSS) | 8 weeks
  A self-administered scale designed to assess nighttime sleep problems, sleep disorders and excessive daytime sleep. Consists of 15 items represented by a ruler (10 cm) where the patient indicates the frequency of the symptom from 0 (always)- 10 (never).

CONTACTS AND LOCATIONS:
Overall Officials: NADJA ASANO, PHD, Principal Investigator — Universidade Federal de Pernambuco